CLINICAL TRIAL: NCT01767415
Title: Intra-operative Use of Indigo Carmine Dye for the Delineation of Ill Defined Tumor Borders Using Stereotactic Injection
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1106011772
Record Dates: First submitted 2013-01-10; First posted 2013-01-14 (Estimated); Results first posted 2018-12-11 (Actual); Last update posted 2018-12-11 (Actual); Status verified 2018-11

CONDITIONS: Brain Tumors With Ill-defined Margins
Keywords: brain tumor; resection; indigo carmine dye
MeSH Terms: conditions — Brain Neoplasms | interventions — Indigo Carmine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Indigo Carmine (Experimental): Intraoperative stereotactic injection of Indigo Carmine
  Interventions: Drug: Indigo carmine

INTERVENTIONS:
Drug: Indigo carmine — During resection, a small quantity of a special dye called indigo carmine will be infused at the margins of the tumor using computer-guided stereotactic navigation equipment. This dye will be visible during the tumor resection and it can potentially serve as an additional marker of the tumor margins. A post-operative MRI scan -which is part of the standard care- will accurately measure the extent of tumor resection.
  Other Names: Indigotindisulfonate sodium

SUMMARY:
The purpose of this study is to investigate whether stereotactic indigo carmine injection can safely increase the extent of tumor resection.

DETAILED DESCRIPTION:
Low grade gliomas are brain tumors with usually poorly defined borders between tumor and normal brain. This characteristic of low grade gliomas makes the gross total resection of the tumor extremely difficult. Nevertheless, several studies have demonstrated that the risk of recurrence and progression into a more malignant tumor can be decreased with a more aggressive surgical resection. An aggressive attempt to achieve a gross total resection may result in the resection of normal brain and therefore neurological injury. For this reason, the more common error is to subtotally resect the tumor leaving significant volumes of tumor behind. Many techniques have been introduced to safely increase the extent of resection, since the extent of resection is associated with a higher survival rate. Each one of these techniques has several shortcomings. The current study will assess whether the intraoperative stereotactic injection of the indigo carmine at the tumor margins helps to safely increase of extent of tumor resection. In the first step of the study the safety and the correlation between resection of stained tissue/extend of tumor resection will be assessed. If the results are satisfactory, then the second step will ensue. In the second step we will assess the utility of indigo carmine as an additional adjunct to guide tumor resection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with gliomas or other tumors that may have ill defined margins during the operative resection.

Exclusion Criteria:

* Subjects with a contraindication for brain MRI scan. Subjects who are pregnant, younger than 18 years old or have a contraindication for indigo carmine are excluded as well

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2012-04 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theodore Schwartz, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medical College Department of Neurological Surgery, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Indigo Carmine
Started | 10
Completed | 10
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Information collected from all study participants.
Arm/Group | Indigo Carmine
Number analyzed (Participants) | 10
Age, Continuous [Mean (Full Range); unit: years] | 49 [25 to 74]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 10
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 10
Region of Enrollment [Number; unit: participants]
  United States | 10
Tumor Location [Count of Participants; unit: Participants]
  Lt Temporal | 1
  Lt Frontal | 2
  Rt frontal | 2
  Lt Occipital | 2
  Rt parietal | 1
  Rt occipital | 1
  Lt parietal | 1
Tumor Diagnosis [Count of Participants; unit: Participants]
  Incidental finding | 3
  Recurrent Disease | 3
  Seizures | 1
  Headache | 1
  Neurological Defect | 2

OUTCOME MEASURES:

1. Primary Outcome: Extent of Resection
Description: Evaluation of the extent of resection of the tumor following the indigo carmine infusion to the tumor.
Time Frame: 48 hours
Population: intraoperative stereotactic injection of indigo carmine at the tumor margins
Measure: Mean (Full Range); unit: percentage of tumor resected
Arm/Group | Indigo Carmine
Number analyzed (Participants) | 10
percentage of tumor resected | 97.1 [91 to 100]

2. Secondary Outcome: Absence of Complications After Injection
Description: Assessment of Post-operative Clinical Course & Complications
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Indigo Carmine
Number analyzed (Participants) | 10
Participants
  Infection | 1
  Hempiaresis | 1
  Mild Word-finding difficulties | 1
  No complications (good clinical course) | 7

ADVERSE EVENTS:
Arm/Group | Indigo Carmine
Serious Adverse Events (participants affected / at risk) | 1/10
Other Adverse Events (participants affected / at risk) | 1/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indigo Carmine (N=10)
Staphylococcus aureus infection (brain abscess) (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Indigo Carmine (N=10)
hemiparesis (Nervous system disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes